CLINICAL TRIAL: NCT05610280
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 3 Study of Olezarsen (ISIS 678354) in Patients With Hypertriglyceridemia and Atherosclerotic Cardiovascular Disease (Established or at Increased Risk for), or With Severe Hypertriglyceridemia
Brief Title: A Study of Olezarsen (ISIS 678354) in Participants With Hypertriglyceridemia and Atherosclerotic Cardiovascular Disease, or With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 678354-CS9; 2022-501486-53 (EudraCT Number)
Expanded Access: NCT06360237 (Approved for marketing)
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hypertriglyceridemia; Cardiovascular Diseases; Atherosclerosis
Keywords: ISIS 678354; Olezarsen
MeSH Terms: conditions — Hypertriglyceridemia; Cardiovascular Diseases; Atherosclerosis | interventions — olezarsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olezarsen (Experimental): Participants will be randomized to receive multiple doses of olezarsen, once every 4 weeks by subcutaneous (SC) injection up to Week 49.
  Interventions: Drug: Olezarsen
- Placebo (Placebo Comparator): Participants will be randomized to receive olezarsen-matching placebo, once every 4 weeks by SC injection up to Week 49.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olezarsen — Olezarsen will be administered by SC injection.
  Other Names: ISIS 678354; AKCEA-APOCIII-LRx
  Arms: Olezarsen
Drug: Placebo — Olezarsen-matching placebo will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of olezarsen on percent change in fasting triglyceride (TG) levels compared to placebo in participants with hypertriglyceridemia and atherosclerotic cardiovascular disease, or with severe hypertriglyceridemia.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, placebo-controlled study in approximately 1475 participants with hypertriglyceridemia and atherosclerotic cardiovascular disease. The study consists of 3 periods: 1) Screening Period: Week -12 to Week -1 (up to 12 weeks); 2) Treatment Period up to Week 53; and 3) Post-Treatment Follow-up Period: Week 54 to Week 66 (13 weeks). Participants enrolled will receive olezarsen or placebo once every 4 weeks during the 53-week Treatment Period.

The Screening Period was extended with no impact to overall study timelines.

A coronary computed tomographic angiography (CTA) sub study will be performed to assess whether triglyceride lowering through inhibition of apoC-III protein synthesis may reduce coronary plaque progression.

ELIGIBILITY:
Inclusion Criteria:

* Participants must fall into 1 of the following groups (a or b):

  a. Hypertriglyceridemia with fasting TG ≥200 mg/dL (2.26 millimoles per liter [mmol/L]) and <500 mg/dL (5.65 mmol/L) with either
* Clinical diagnosis of atherosclerotic cardiovascular disease (ASCVD) or
* At increased risk for ASCVD

  b. Severe hypertriglyceridemia with fasting TG ≥500 mg/dL (5.65 mmol/L)
* Participants should be on standard of care (SOC) lipid-lowering medications per local guidelines. Lipid-lowering medications should be optimized and stabilized for at least 4 weeks prior to Screening to minimize changes in these medications during the study.

Exclusion Criteria:

* Hemoglobin A1c (HbA1c) ≥ 9.5% at Screening
* Alanine aminotransferase or aspartate aminotransferase > 3.0 × upper limit of normal
* Total bilirubin > 1.5 upper limit of normal unless due to Gilbert's syndrome
* Estimated GFR < 30 mL/min/1.73 m^2

NOTE: Other Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1478 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline to Week 25 in Fasting Triglycerides (TG) Compared to Placebo | Baseline to Week 25

SECONDARY OUTCOMES:
Percent Change From Baseline to Week 53 in Fasting TG Compared to Placebo | Baseline to Week 53
Proportion of Participants who Achieve Fasting TG <150 Milligrams per Deciliter (mg/dL) at Weeks 25 and 53 Compared to Placebo | Baseline, Weeks 25 and 53
Percent Change From Baseline to Weeks 25 and 53 in Fasting Apolipoprotein C-III (apoC-III) Compared to Placebo | Baseline to Weeks 25 and 53
Percent Change From Baseline to Weeks 25 and 53 in Fasting Very Low-Density Lipoprotein-Cholesterol (VLDL)-C Compared to Placebo | Baseline to Weeks 25 and 53
Percent Change From Baseline to Weeks 25 and 53 in Fasting Remnant Cholesterol Compared to Placebo | Baseline to Weeks 25 and 53
Percent Change From Baseline to Weeks 25 and 53 in Fasting non-High Density Lipoprotein-Cholesterol (HDL)-C Compared to Placebo | Baseline to Weeks 25 and 53
Percent Change From Baseline to Weeks 25 and 53 in Fasting High-Density Lipoprotein-Cholesterol (HDL)-C Compared to Placebo | Baseline to Weeks 25 and 53
Percent Change From Baseline to Weeks 25 and 53 in Fasting Apolipoprotein B (apoB) Compared to Placebo | Baseline to Weeks 25 and 53
Percent Change From Baseline to Weeks 25 and 53 in Fasting Low-Density Lipoprotein-Cholesterol (LDL)-C Compared to Placebo | Baseline to Weeks 25 and 53

CONTACTS AND LOCATIONS:
Locations (167):
- United States (67):
  - Alabama Clinical Therapeutics, LLC Alabaster, Birmingham, Alabama
  - Heart Center Research PC, Huntsville, Alabama
  - Cardiovascular Research Foundation of Southern California, Beverly Hills, California
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - Diabetes/Lipid Management & Research Center, Huntington Beach, California
  - University of California, San Diego (UCSD), La Jolla, California
  - Clinical Trials Research, Lincoln, California
  - Amicis Research, Northridge, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Northern California Research, Sacramento, California
  - Amicis Research Center, Santa Clarita, California
  - Metabolic Institute of America, Tarzana, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California
  - Amicis Research Center, Valencia, California
  - Excel Clinical Medical Trials, Boca Raton, Florida
  - Finlay Medical Research - West Palm, Greenacres City, Florida
  - Global Research Associates, Homestead, Florida
  - 3Sync Research, Lake Worth, Florida
  - Finlay Medical Research, Miami, Florida
  - Advanced Medical Research Institute (AMRI), Miami, Florida
  - De La Cruz Research Center, LL, Miami, Florida
  - Suncoast Clinical Research, Inc. - New Port Richey, New Port Richey, Florida
  - Suncoast Clinical Research, Inc. - Palm Harbor, New Port Richey, Florida
  - Proactive Clinical Research, Oakland Park, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Comprehensive Medical & Research Center, Plantation, Florida
  - Progressive Medical Research, Port Orange, Florida
  - St. Johns Center for Clinical Research, Saint Augustine, Florida
  - JSV Clinical Research Study, Inc, Tampa, Florida
  - Centricity Research, Columbus, Georgia
  - Atlanta Heart Specialists, Tucker, Georgia
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - Affinity Health, Park Ridge, Illinois
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Mercy One Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - Norton Cardiovascular Associates, Louisville, Kentucky
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Aa Mrc, Llc, Flint, Michigan
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Medical University of South Carolina (MUSC), Charleston, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Aultman Hospital Cardiology Clinical Trials, Canton, Ohio
  - McConnell Heart Health Center, Columbus, Ohio
  - Summit Research Group, LLC, Stow, Ohio
  - Central Oklahoma Early Detection Center, Edmond, Oklahoma
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Main Street Physicians Care Waterway, Little River, South Carolina
  - OnSite Clinical Solutions, LLC, Rock Hill, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Health Concepts, Rapid City, South Dakota
  - The Jackson Clinic, Jackson, Tennessee
  - Affinity Health Corp., Nashville, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - FMC Science, Round Rock, Texas
  - Carient Heart & Vascular, Manassas, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Charleston Area Medical Center (CAMC) Clinical Trials Center, Charleston, West Virginia
- Bulgaria (11):
  - MHAT Sv. Ivan Rilski - 2003 OOD, Dupnitsa
  - University Multiprofile Hospital for Active Treatment Pulmed OOD, Plovdiv
  - SHATC Medica Cor EAD, Rousse
  - Medical Center for Specialized Medical Help in Cardiovascular Diseases OOD, Sofia
  - MBAL National Cardiology Hospital, Sofia
  - University Multiprofile Hospital for Active Treatment Alexandrovska, Sofia
  - University Multiprofile Hospital for Active Treatment, Sofia
  - Medico Dental Center ISUL Tsaritsa Yoanna EOOD, Sofia
  - UMHAT Prof. Dr. Stoyan Kirkovich, Stara Zagora
  - Diagnostic Consultative Center Equita (DCC Equita), Varna
  - Specialized Hospital for Active Treatment of Cardiology, Varna
- Canada (13):
  - ARC Biosystems, Vancouver, British Columbia
  - Centricity Research - Vaughan Endocrinology, Concord, Ontario
  - Centricity Research - Etobicoke Endocrinology, Etobicoke, Ontario
  - Centricity Research - Oshawa Multispecialty, Oshawa, Ontario
  - Bluewater Clinical Research Group Inc, Sarnia, Ontario
  - Centricity Research - Toronto LMC Multispecialty, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Montreal Heart Institute - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Institute de Recherches Cliniques de Montreal, Montreal, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec, Quebec
  - Centricity Research - Barrie Endocrinology, Barrie
  - Centricity Research - Brampton Endocrinology, Brampton
  - Centre de Recherche Saint-Louis, Québec
- Czechia (8):
  - UNIVMED s.r.o. - Kardiologicka Ambulance, Brno
  - Cevni ambulance - MATMED s.r.o., Hodonín
  - Edumed s.r.o., Kardiologicka, endokrinologicka, diabetologicka a interni ambulance Nachod, Jaroměř
  - Affidea Praha s.r.o., Prague
  - Diabetologicka a endokrinologicka ambulance Milan Kvapil s.r.o, Prague
  - Endokrinologie Cerny Most s.r.o., Prague
  - AeskuLab k.s, Teplice
  - MUDr. Nina Zemkova s.r.o. Interni Ambulance, Uherské Hradiště
- Denmark (6):
  - Aarhus University Hospital, Aarhus
  - Sydvestjysk Hospital, Esbjerg
  - Gentofte Hospital, Hellerup
  - Godstrup Regional Hospital (Gødstrup), Herning
  - OUH Svendborg Hospital, Svendborg
  - Viborg Regional Hospital, Viborg
- France (5):
  - HCL Hopital Louis Pradel, Bron
  - CHU Dijon Bourgogne - Hopital Francois Mitterrand, Dijon
  - AP-HP Hopital Pitie-Salpetriere, Paris
  - Groupement de Cooperation Sanitaire (GCS) ELSAN - Polyclinique Vauban, Valenciennes
  - GHM les Portes du Sud, Vénissieux
- Hungary (3):
  - Clinexpert Kft., Budapest
  - Obudai Egeszsegugyi Centrum, Budapest
  - CRU Hungary Kft., Encs
- Italy (7):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - ASST NORD MILANO-Ospedale Edoardo Bassini, Cinisello Balsamo
  - Azienda Ospedaliero-Universitaria di Ferrara-Arcispedale Sant'Anna, Cona
  - Centro Cardiologico Monzino, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
- Netherlands (15):
  - Academic Medical Center - Department of Vascular Medicine, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Het Van Weel-Bethesda Ziekenhuis, Dirksland
  - Groene Hart Ziekenhuis, Gouda
  - Spaarne Gasthuis, Haarlem
  - Zuyderland Medisch Centrum, Heerlen
  - Bethesda Diabetes Research Center, Hoogeveen
  - Canisius-Wilhelmina Ziekenhuis (CWZ), Nijmegen
  - D&A Research, Sneek
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - Albert Schweitzer Ziekenhuis - Location Dordrecht, Zwijndrecht
  - Albert Schweitzer Ziekenhuis, Zwijndrecht
- The Lipid Clinic (Oslo University Hospital), Oslo, Norway
- Poland (13):
  - SALVIA Lekston i Madej s.j., Katowice
  - Jagiellonskie Centrum Innowacji Sp. z o.o., Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - FutureMeds, Lodz
  - INSTYTUT CENTRUM ZDROWIA MATKI POLKI - Klinika Kardiologii i Wad Wrodzonych Doroslych, Lodz
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - FutureMeds Warszawa Centrum, Warsaw
  - Clinical Best Solutions Sp. z.o.o Spolka Komandytowa, Warsaw
  - FutureMeds - Centrum Medyczne AMED Warszawa Targowek, Warsaw
  - Narodowy Instytut Kardiologii Stefana kardynala Wyszynskiego - Panstwowy Instytut Badawczy, Klinika Kardiologii i Angiologii Interwencyjnej, Warsaw
  - FutureMeds Sp. z o.o, Wroclaw
  - Slaski Park Technologii Medycznych Kardio-Med Silesia Sp. z o. o, Zabrze
  - ETG Zamosc - Pro Life Medica Sp. z o.o, Zamość
- Portugal (4):
  - Centro Hospitalar de Lisboa Ocidental. E.P.E, - Hospital Santa Cruz, Carnaxide
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - Centro Hospitalar Universitario de Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia/Espinho EPE, Vila Nova de Gaia
- Slovakia (4):
  - Alian, s.r.o., Kardiologicka ambulancia, Bardejov
  - Cardio D&R, S.R.O. Kosice, Košice
  - Diab sro, Rožňava
  - Interna SK, s.r.o., Kardiologicka a interna ambulancia, Svidník
- Spain (10):
  - Hospital Abente y Lago, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Calle Villarroel 170, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/

REFERENCES:
- [Derived] Bergmark BA, Marston NA, Prohaska TA, Alexander VJ, Zimerman A, Moura FA, Kang YM, Weinland J, Murphy SA, Goodrich EL, Zhang S, Li D, Banach M, Stroes E, Lu MT, Tsimikas S, Giugliano RP, Sabatine MS; Essence-TIMI 73b Investigators. Targeting APOC3 with Olezarsen in Moderate Hypertriglyceridemia. N Engl J Med. 2025 Oct 2;393(13):1279-1291. doi: 10.1056/NEJMoa2507227. Epub 2025 Aug 30. PMID 40888739
- [Derived] Bergmark BA, Marston NA, Prohaska TA, Alexander VJ, Zimerman A, Moura FA, Kang YM, Murphy SA, Zhang S, Lu MT, Karwatowska-Prokopczuk E, Tsimikas S, Giugliano RP, Sabatine MS. Olezarsen in patients with hypertriglyceridemia at high cardiovascular risk: Rationale and design of the Essence-TIMI 73b trial. Am Heart J. 2025 Aug;286:116-124. doi: 10.1016/j.ahj.2025.02.022. Epub 2025 Mar 11. PMID 40081744